## Development of methods and algorithms for diet design based on gut microbiota analysis

## **Consent letter**

Number of clinical trial: 1631 Project number: NSP67

Approved by Ethical Committe of National Institute for Health Development 25.10.2016

## Consent to be involved in the study: Development of methods and algorithms for diet design based on gut microbiota analysis

I have been informed that my participation in this study is voluntary. I may terminate my participation in the study at any time without giving reasons for my decision. Refusal to participate or subsequent withdrawal will not have any negative consequences for me.

I have read the aims of the study and the content of the study has been explained to me. I agree to the processing of all non-personal data collected about me during the study, both at the Institute for Health Development and within the project by its contractual partners. Data collected about me may only be published in a non-personalized form. If I have any additional questions, I know who I can contact from the Institute for Health Development.

I confirm that I have not been diagnosed with long-term or chronic diseases or symptoms and that I have no restrictions on food choices (allergies, food intolerances, vegetarianism, etc.). In addition, I confirm that I have not used antibiotics in the last three months and have not traveled to subtropical or tropical regions in the last one month.

I agree to participate in the study "Development of methods and algorithms for diet design based on gut microbiota analysis" and to the processing of the study data in accordance with the personal data protection Law and I confirm this with my signature.

| Participant name: |
|---|
| Contacts: |
| □ I would like to receive sample collection tools within a business day at: |
| □ I would like to receive sample collection equipment at the Omniva parcel machine, write down the exact name of the parcel machine: |
| Phone: e-mail: |
| E-mail and phone are used only to transmit survey-related information. |
| I would like to answer questionnaire: □ on the web. □ in the file. □ on the paper. |
| I would like feedback on my research findings and dietary recommendations. □ via encrypted e-mail. □ via registered mail. |
| □ I do not want feedback on my research results. |
| (digitally signed) |